CLINICAL TRIAL: NCT01764451
Title: Permeability MRI in Cerebral Cavernous Malformations Type 1 in New Mexico: Effects of Statins
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Research was completed before January 18, 2017, & does not meet the Applicable Clinical Trial requirement to register & report results per the guidance provided in "Clinical Trials Registration & Results Information Submission" dated 09/21/2016.
Sponsor: University of New Mexico (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Leslie Morrison, Vice Chancellor for Academic Affairs, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BVMC 6205; U54NS065705 (NIH)
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cavernous Angioma, Familial; Cerebral Cavernous Malformations; Cerebral Cavernous Hemangioma
Keywords: Hispanic
MeSH Terms: conditions — Hemangioma, Cavernous, Central Nervous System | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin (Experimental): 20-40 mg tablet taken daily by mouth. Month 1: 20 mg; Months 2 and 3: 40 mg.
  Interventions: Drug: Simvastatin
- No Treatment (No Intervention)

INTERVENTIONS:
Drug: Simvastatin
  Other Names: Zocor
  Arms: Simvastatin

SUMMARY:
Cerebral cavernous malformations (CCMs) are clusters of abnormal blood vessels in the brain and spine. CCMs can bleed and cause strokes, seizures, and headaches. In some patients, CCMs affect the blood brain barrier (BBB). The BBB is the body's separation of blood and its contents in the brain from the brain tissue itself. Abnormal leakiness or permeability of this barrier can cause disease. We will measure the permeability (leakiness) of the BBB using a magnetic resonance imaging (MRI) technique called dynamic contrast-enhanced MRI (DCEMRI). The purpose of this study is to look at whether statin medications change the permeability (leakiness) of the blood brain barrier in CCM patients. Statin medications are used to lower cholesterol levels and prevent heart attack and stroke. In addition, this medication may decrease the risk of brain hemorrhage or bleeding in patients with CCM. This study will examine whether the permeability of the BBB changes following the administration of simvastatin for three months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral cavernous malformations-common Hispanic mutation (CCM1-CHM)
* Must be willing to travel to the University of New Mexico in Albuquerque, NM for 5 visits over the course of three months.

Exclusion Criteria:

* Incarceration
* Unable to pass MRI safety screening (pregnant females, claustrophics, or those with certain metallic items implanted in their bodies)
* Low kidney function or transplants, an eGFR below 60 mL/min
* Currently taking statin medications or have taken statin medications in the past 6 months
* Known allergy or intolerance to statins
* Known allergy or intolerance to gadolinium
* Liver dysfunction at baseline, AST > 47 and/or ALT > 49
* Consumption of large quantities of alcohol, men who consume more than 2 daily drinks and women who consume more than one daily drink
* CK level of 232 or higher
* Triglycerides greater than or equal to 500.
* Medications: gemfibrozil, cyclosporine, danazol, itraconazole, ketoconazole, posaconazole, ethromycin, clarithomycin, telithromycin, HIV protease inhibitors, nefazoldone, amiodarone, verapamil, dilitiazem, amlodipine, or ranalazine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in blood brain barrier permeability over three months for the treatment group compared to the control group. | Baseline, Three Months
  We will measure the change in blood brain barrier permeability with dynamic contrast enhanced MRI from baseline to three months. We will compare the change in permeability for a group of CCM patients placed on statin medication (treatment group) with a group of CCM patients not on statin medication (control group).

SECONDARY OUTCOMES:
Correlation of physiologic permeability data with anatomic lesion data | Baseline, Three months
  Use dynamic contrast-enhanced MRI to detect abnormalities in brain permeability in CCM patients and correlate with anatomic lesion information.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A Morrison, MD, Principal Investigator — University of New Mexico; Blaine Hart, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

REFERENCES:
- See also: Angioma Alliance is an organization by and for those affected by cavernous angiomas and their loved ones, health professionals, and researchers. — http://www.angiomaalliance.org/